CLINICAL TRIAL: NCT04590937
Title: The Effect of BI 730357 on the Pharmacokinetics of Rosuvastatin, Digoxin, Metformin and Furosemide Given as a Cocktail - an Open-label, Non-randomised, 2-period Fixed-sequence Trial in Healthy Subjects
Brief Title: A Study in Healthy People to Test Whether BI 730357 Affects How 4 Other Medicines (Rosuvastatin, Digoxin, Metformin, and Furosemide) Are Taken up in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1407-0038; 2020-003097-46 (EudraCT Number)
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; Digoxin; Metformin; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cocktail/ Cocktail + BI 730357 (Experimental): Cocktail treatment will be followed by the Test treatment in a fixed sequence. The treatment periods are separated by a wash-out phase of at least 14 days between the two cocktail administrations.
  Interventions: Drug: BI 730357; Drug: CRESTOR®; Drug: Lenoxin®; Drug: MetfoLiquid GeriaSan®; Drug: Lasix®

INTERVENTIONS:
Drug: BI 730357 — Film-coated tablet
Drug: CRESTOR® — Film-coated tablet
  Other Names: Rosuvastatin
Drug: Lenoxin® — Tablet
  Other Names: Digoxin
Drug: MetfoLiquid GeriaSan® — Oral solution
  Other Names: Metformin hydrochloride
Drug: Lasix® — Oral solution
  Other Names: Furosemide

SUMMARY:
The main objective of this trial is to investigate the effect of BI 730357 under steady state conditions on the pharmacokinetics of digoxin, furosemide, metformin and rosuvastatin given as a cocktail (Reference, R: cocktail alone; Test T: cocktail given under steady state conditions of BI 730357).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory Tests
* Age of 18 to 55 years (inclusive)
* BMI of 18.5 to 29.9 kilogram per square meter (kg/m2) (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects, or female subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion: -- Use of adequate contraception, e.g. any of the following methods plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device

  * Sexually abstinent
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy or bilateral tubal occlusion)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with levels of Follicle-stimulating hormone (FSH) above 40 units per liter (U/L) and estradiol below 30 nanograms per liter (ng/L) is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetres of Mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* During COVID-19 pandemic: laboratory test indicative of an ongoing SARS-CoV-2 infection
* further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label, non-randomised, 2-period fixed-sequence trial in healthy subjects was to test whether BI 730357 affects how 4 other medicines (rosuvastatin, digoxin, metformin, and furosemide) are taken up in the body.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Cocktail (R) / BI 730357+Cocktail (T): Each subject participated in 2 treatment periods (Days -1 to 7 in period 1 and Days -7 to Day 8 in Period 2).
  In period 1 (Visit 2): the cocktail reference treatment (R) consisting of 1 tablet of 0.25 milligrams (mg) of Digoxin, 0.1 milliliter (mL) oral solution of 1 mg Furosemide, 0.05 mL oral solution of 10 mg Metformin, and 1 film-coated tablet of 10 mg Rosuvastatin were taken orally, each medication as a single dose, once on Day 1 of period 1 (Visit 2).
  In period 2 (Visit 3): 3 film-coated tablets of 100 mg BI 730357 were taken orally twice daily (bid) (daily dose 600 mg) from Day -7 until Day 6 of Visit 3 (13 days in total). On Day 1 of Visit 3, 1 hour after the morning dose of BI 730357, the cocktail (1 tablet of 0.25 mg of Digoxin, 0.1 mL oral solution of 1 mg Furosemide, 0.05 mL oral solution of 10 mg Metformin, and 1 film-coated tablet of 10 mg Rosuvastatin) was administered orally once. The BI 730357+ cocktail was the test treatment (T).
  The two cocktail administrations were separated by a wash-out period of at least 14 days.
Period: Period 1 - Cocktail
Arm/Group | Cocktail (R) / BI 730357+Cocktail (T)
Started | 15
Completed ("completed" refers to: not prematurely discontinued from trial medication) | 15
Not Completed | 0
Period: Period 2 - BI 730357+Cocktail
Arm/Group | Cocktail (R) / BI 730357+Cocktail (T)
Started | 15
Treated at Least One Dose of BI | 15
Treated at Least One Dose of Cocktail+BI | 14
Completed ("completed" refers to: not prematurely discontinued from trial medication) | 14
Not Completed | 1
Not completed — COVID-19 related | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set includes all subjects who signed informed consent and were treated with at least one dose of study drug.
Arm/Group | Cocktail (R) / BI 730357+Cocktail (T)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Metformin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞, Metformin)
Description: Area under the concentration-time curve of Metformin in plasma over the time interval from 0 extrapolated to infinity is reported. The geometric mean is actually adjusted geometric mean.
Time Frame: 2 hours (h) before and at 20 minutes (min), 40min, 1h, 1h30min, 2h, 2h30min, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 71h, 95h after administration of Metformin in both periods plus at 143h in period 1 and at 119h and 167h in period 2.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set includes all subjects in the Treated Set who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject is included in the PKS, even if he/she contributes only one PK parameter value for one period to the statistical assessment. Only those with non-missing results are included in the analysis.
Measure: Geometric Mean (Standard Error); unit: hour * nanomole / liter (h*nmol/L)
Groups:
- Metformin (Period 1): In period 1 (Visit 2): 0.05 milliliter (mL) oral solution of 10 milligrams (mg) Metformin were taken orally as a single dose once on Day 1 of period 1 (Visit 2).
- Metformin + BI 730357 (Period 2): In period 2 (Visit 3): 3 film-coated tablets of 100 mg BI 730357 were taken orally twice daily (bid) with daily dose 600 mg from Day -7 until Day 6 of Visit 3 (13 days in total). On Day 1 of Visit 3, 1 hour after the morning dose of BI 730357, 0.05 mL oral solution of 10 mg Metformin were administered orally once. The two Metformin administrations were separated by a wash-out period of at least 14 days.
Arm/Group | Metformin (Period 1) | Metformin + BI 730357 (Period 2)
Number analyzed (Participants) | 15 | 14
hour * nanomole / liter (h*nmol/L) | 1460.83 (NA) — Standard Error is adjusted geometric Standard Error = 1.05 | 1434.81 (NA) — Standard Error is adjusted geometric Standard Error = 1.05
Statistical Analysis 1: Comparison: Metformin (Period 1) vs Metformin + BI 730357 (Period 2); Test type: Other — ANOVA model including "subject" as random and "treatment" as fixed effect was used; Geometric means ratio = 98.22, 90% CI 2-sided [94.89 to 101.67], Standard Error of Mean 5.2 — The geometric means ratio was calculated as Metformin + BI 730357 / Metformin. Standard error of the mean is actually the intra-individual geometric coefficient of variation (gCV)

2. Primary Outcome: Area Under the Concentration-time Curve of Rosuvastatin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞, Rosuvastatin)
Description: Area under the concentration-time curve of Rosuvastatin in plasma over the time interval from 0 extrapolated to infinity is reported. The geometric mean is actually adjusted geometric mean.
Time Frame: 2 hours (h) before and at 20 minutes (min), 40min, 1h, 1h30min, 2h, 2h30min, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 71h, 95h after administration of Rosuvastatin in both periods plus at 143h in period 1 and at 119h and 167h in period 2.
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: hour * nanomole / liter (h*nmol/L)
Groups:
- Rosuvastatin (Period 1): In period 1 (Visit 2): 1 film-coated tablet of 10 milligrams (mg) Rosuvastatin was taken orally as a single dose once on Day 1 of period 1 (Visit 2).
- Rosuvastatin + BI 730357 (Period 2): In period 2 (Visit 3): 3 film-coated tablets of 100 mg BI 730357 were taken orally twice daily (bid) with daily dose 600 mg from Day -7 until Day 6 of Visit 3 (13 days in total). On Day 1 of Visit 3, 1 hour after the morning dose of BI 730357, 1 film-coated tablet of 10 mg Rosuvastatin was administered orally once. The two Rosuvastatin administrations were separated by a wash-out period of at least 14 days.
Arm/Group | Rosuvastatin (Period 1) | Rosuvastatin + BI 730357 (Period 2)
Number analyzed (Participants) | 14 | 13
hour * nanomole / liter (h*nmol/L) | 90.08 (NA) — Standard Error is adjusted geometric Standard Error = 1.11 | 110.87 (NA) — Standard Error is adjusted geometric Standard Error = 1.12
Statistical Analysis 1: Comparison: Rosuvastatin (Period 1) vs Rosuvastatin + BI 730357 (Period 2); Test type: Other — ANOVA model including "subject" as random and "treatment" as fixed effect was used; Geometric means ratio = 123.08, 90% CI 2-sided [112.22 to 134.98], Standard Error of Mean 12.7 — The geometric means ratio was calculated as Rosuvastatin + BI 730357 / Rosuvastatin. Standard error of the mean is actually the intra-individual geometric coefficient of variation (gCV)

3. Primary Outcome: Area Under the Concentration-time Curve of Furosemide in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞, Furosemide)
Description: Area under the concentration-time curve of Furosemide in plasma over the time interval from 0 extrapolated to infinity is reported. The geometric mean is actually adjusted geometric mean.
Time Frame: 2 hours (h) before and at 20 minutes (min), 40min, 1h, 1h30min, 2h, 2h30min, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 71h, 95h after administration of Furosemide in both periods plus at 143h in period 1 and at 119h and 167h in period 2.
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: hour * nanomole / liter (h*nmol/L)
Groups:
- Furosemide (Period 1): In period 1 (Visit 2): 0.1 milliliter (mL) oral solution of 1 milligrams (mg) Furosemide were taken orally as a single dose once on Day 1 of period 1 (Visit 2).
- Furosemide + BI 730357 (Period 2): In period 2 (Visit 3): 3 film-coated tablets of 100 mg BI 730357 were taken orally twice daily (bid) with daily dose 600 mg from Day -7 until Day 6 of Visit 3 (13 days in total). On Day 1 of Visit 3, 1 hour after the morning dose of BI 730357, 0.1 milliliter (mL) oral solution of 1 milligrams (mg) Furosemide were administered orally once. The two Furosemide administrations were separated by a wash-out period of at least 14 days.
Arm/Group | Furosemide (Period 1) | Furosemide + BI 730357 (Period 2)
Number analyzed (Participants) | 15 | 13
hour * nanomole / liter (h*nmol/L) | 157.57 (NA) — Standard Error is adjusted geometric Standard Error = 1.06 | 185.50 (NA) — Standard Error is adjusted geometric Standard Error = 1.06
Statistical Analysis 1: Comparison: Furosemide (Period 1) vs Furosemide + BI 730357 (Period 2); Test type: Other — ANOVA model including "subject" as random and "treatment" as fixed effect was used; Geometric means ratio = 117.72, 90% CI 2-sided [110.57 to 125.34], Standard Error of Mean 9.0 — The geometric means ratio was calculated as Furosemide + BI 730357 / Furosemide. Standard error of the mean is actually the intra-individual geometric coefficient of variation (gCV)

4. Primary Outcome: Area Under the Concentration-time Curve of Digoxin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞, Digoxin)
Description: Area under the concentration-time curve of Digoxin in plasma over the time interval from 0 extrapolated to infinity is reported. The geometric mean is actually adjusted geometric mean.
Time Frame: 2 hours (h) before and at 20 minutes (min), 40min, 1h, 1h30min, 2h, 2h30min, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 71h, 95h after administration of Digoxin in both periods plus at 143h in period 1 and at 119h and 167h in period 2.
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: hour * nanomole / liter (h*nmol/L)
Groups:
- Digoxin (Period 1): In period 1 (Visit 2): 1 tablet of 0.25 milligrams (mg) of Digoxin was taken orally as a single dose once on Day 1 of period 1 (Visit 2).
- Digoxin + BI 730357 (Period 2): In period 2 (Visit 3): 3 film-coated tablets of 100 mg BI 730357 were taken orally twice daily (bid) with daily dose 600 mg from Day -7 until Day 6 of Visit 3 (13 days in total). On Day 1 of Visit 3, 1 hour after the morning dose of BI 730357, 1 tablet of 0.25 mg Digoxin was administered orally once. The two Digoxin administrations were separated by a wash-out period of at least 14 days.
Arm/Group | Digoxin (Period 1) | Digoxin + BI 730357 (Period 2)
Number analyzed (Participants) | 15 | 14
hour * nanomole / liter (h*nmol/L) | 13.34 (NA) — Standard Error is adjusted geometric Standard Error = 1.09 | 22.71 (NA) — Standard Error is adjusted geometric Standard Error = 1.10
Statistical Analysis 1: Comparison: Digoxin (Period 1) vs Digoxin + BI 730357 (Period 2); Test type: Other — ANOVA model including "subject" as random and "treatment" as fixed effect was used; Geometric means ratio = 170.29, 90% CI 2-sided [143.73 to 201.76], Standard Error of Mean 25.6 — The geometric means ratio was calculated as Digoxin + BI 730357 / Digoxin. Standard error of the mean is actually the intra-individual geometric coefficient of variation (gCV)

5. Primary Outcome: Maximum Measured Concentration of Metformin in Plasma (Cmax, Metformin)
Description: Maximum measured concentration of Metformin in plasma is reported. The geometric mean is actually adjusted geometric mean.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomole / liter (nmol/L)
Arm/Group | Metformin (Period 1) | Metformin + BI 730357 (Period 2)
Number analyzed (Participants) | 15 | 14
nanomole / liter (nmol/L) | 235.86 (NA) — Standard Error is adjusted geometric Standard Error = 1.04 | 215.63 (NA) — Standard Error is adjusted geometric Standard Error = 1.04
Statistical Analysis 1: Comparison: Metformin (Period 1) vs Metformin + BI 730357 (Period 2); Test type: Other — ANOVA model including "subject" as random and "treatment" as fixed effect was used; Geometric means ratio = 91.42, 90% CI 2-sided [88.04 to 94.93], Standard Error of Mean 5.6 — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Maximum Measured Concentration of Rosuvastatin in Plasma (Cmax, Rosuvastatin)
Description: Maximum measured concentration of Rosuvastatin in plasma is reported. The geometric mean is actually adjusted geometric mean.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomole / liter (nmol/L)
Arm/Group | Rosuvastatin (Period 1) | Rosuvastatin + BI 730357 (Period 2)
Number analyzed (Participants) | 15 | 14
nanomole / liter (nmol/L) | 6.92 (NA) — Standard Error is adjusted geometric Standard Error = 1.13 | 9.63 (NA) — Standard Error is adjusted geometric Standard Error = 1.13
Statistical Analysis 1: Comparison: Rosuvastatin (Period 1) vs Rosuvastatin + BI 730357 (Period 2); Test type: Other — ANOVA model including "subject" as random and "treatment" as fixed effect was used; Geometric means ratio = 139.03, 90% CI 2-sided [124.29 to 155.51], Standard Error of Mean 16.9 — [estimate comment as in outcome 2, analysis 1]

7. Primary Outcome: Maximum Measured Concentration of Furosemide in Plasma (Cmax, Furosemide)
Description: Maximum measured concentration of Furosemide in plasma is reported. The geometric mean is actually adjusted geometric mean.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: hour * nanomole / liter (h*nmol/L)
Arm/Group | Furosemide (Period 1) | Furosemide + BI 730357 (Period 2)
Number analyzed (Participants) | 15 | 14
hour * nanomole / liter (h*nmol/L) | 51.03 (NA) — Standard Error is adjusted geometric Standard Error = 1.08 | 57.21 (NA) — Standard Error is adjusted geometric Standard Error = 1.09
Statistical Analysis 1: Comparison: Furosemide (Period 1) vs Furosemide + BI 730357 (Period 2); Test type: Other — ANOVA model including "subject" as random and "treatment" as fixed effect was used; Geometric means ratio = 112.10, 90% CI 2-sided [101.26 to 124.11], Standard Error of Mean 15.4 — [estimate comment as in outcome 3, analysis 1]

8. Primary Outcome: Maximum Measured Concentration of Digoxin in Plasma (Cmax, Digoxin)
Description: Maximum measured concentration of Digoxin in plasma is reported. The geometric mean is actually adjusted geometric mean.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomole / liter (nmol/L)
Arm/Group | Digoxin (Period 1) | Digoxin + BI 730357 (Period 2)
Number analyzed (Participants) | 15 | 14
nanomole / liter (nmol/L) | 0.87 (NA) — Standard Error is adjusted geometric Standard Error = 1.16 | 1.40 (NA) — Standard Error is adjusted geometric Standard Error = 1.16
Statistical Analysis 1: Comparison: Digoxin (Period 1) vs Digoxin + BI 730357 (Period 2); Test type: Other — ANOVA model including "subject" as random and "treatment" as fixed effect was used; Geometric means ratio = 161.29, 90% CI 2-sided [129.17 to 201.39], Standard Error of Mean 34.1 — [estimate comment as in outcome 4, analysis 1]

9. Secondary Outcome: Area Under the Concentration-time Curve of Metformin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz, Metformin)
Description: Area under the concentration-time curve of Metformin in plasma over the time interval from 0 to the last quantifiable data point is reported. The geometric mean is actually adjusted geometric mean.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: hour * nanomole / liter (h*nmol/L)
Arm/Group | Metformin (Period 1) | Metformin + BI 730357 (Period 2)
Number analyzed (Participants) | 15 | 14
hour * nanomole / liter (h*nmol/L) | 1450.30 (NA) — Standard Error is adjusted geometric Standard Error = 1.05 | 1424.70 (NA) — Standard Error is adjusted geometric Standard Error = 1.05
Statistical Analysis 1: Comparison: Metformin (Period 1) vs Metformin + BI 730357 (Period 2); Test type: Other — ANOVA model including "subject" as random and "treatment" as fixed effect was used; Geometric means ratio = 98.23, 90% CI 2-sided [94.86 to 101.73], Standard Error of Mean 5.2 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Area Under the Concentration-time Curve of Rosuvastatin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz, Rosuvastatin)
Description: Area under the concentration-time curve of Rosuvastatin in plasma over the time interval from 0 to the last quantifiable data point is reported. The geometric mean is actually adjusted geometric mean.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: hour * nanomole / liter (h * nmol/L)
Arm/Group | Rosuvastatin (Period 1) | Rosuvastatin + BI 730357 (Period 2)
Number analyzed (Participants) | 15 | 14
hour * nanomole / liter (h * nmol/L) | 78.83 (NA) — Standard Error is adjusted geometric Standard Error = 1.14 | 93.54 (NA) — Standard Error is adjusted geometric Standard Error = 1.14
Statistical Analysis 1: Comparison: Rosuvastatin (Period 1) vs Rosuvastatin + BI 730357 (Period 2); Test type: Other — ANOVA model including "subject" as random and "treatment" as fixed effect was used; Geometric means ratio = 118.67, 90% CI 2-sided [108.83 to 129.40], Standard Error of Mean 13.0 — [estimate comment as in outcome 2, analysis 1]

11. Secondary Outcome: Area Under the Concentration-time Curve of Furosemide in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz, Furosemide)
Description: Area under the concentration-time curve of Furosemide in plasma over the time interval from 0 to the last quantifiable data point is reported. The geometric mean is actually adjusted geometric mean.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: hour * nanomole / liter (h*nmol/L)
Arm/Group | Furosemide (Period 1) | Furosemide + BI 730357 (Period 2)
Number analyzed (Participants) | 15 | 14
hour * nanomole / liter (h*nmol/L) | 151.01 (NA) — Standard Error is adjusted geometric Standard Error = 1.05 | 172.26 (NA) — Standard Error is adjusted geometric Standard Error = 1.06
Statistical Analysis 1: Comparison: Furosemide (Period 1) vs Furosemide + BI 730357 (Period 2); Test type: Other — ANOVA model including "subject" as random and "treatment" as fixed effect was used; Geometric means ratio = 114.07, 90% CI 2-sided [107.93 to 120.56], Standard Error of Mean 8.3 — [estimate comment as in outcome 3, analysis 1]

12. Secondary Outcome: Area Under the Concentration-time Curve of Digoxin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz, Digoxin)
Description: Area under the concentration-time curve of Digoxin in plasma over the time interval from 0 to the last quantifiable data point is reported. The geometric mean is actually adjusted geometric mean.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: hour * nanomole / liter (h*nmol/L)
Arm/Group | Digoxin (Period 1) | Digoxin + BI 730357 (Period 2)
Number analyzed (Participants) | 15 | 14
hour * nanomole / liter (h*nmol/L) | 11.00 (NA) — Standard Error is adjusted geometric Standard Error = 1.10 | 19.11 (NA) — Standard Error is adjusted geometric Standard Error = 1.11
Statistical Analysis 1: Comparison: Digoxin (Period 1) vs Digoxin + BI 730357 (Period 2); Test type: Other — ANOVA model including "subject" as random and "treatment" as fixed effect was used; Geometric means ratio = 173.77, 90% CI 2-sided [141.90 to 212.80], Standard Error of Mean 30.8 — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Cocktail: From 1st dose of cocktail until 1st dose of BI 730357 (BI) or end of 10 days residual effect period (REP) of cocktail, whichever occurs earlier, up to 10 days. Cocktail+BI: the period where the REP of the 1st dose of cocktail overlaps with the start of the dosing of BI, up to 3 days. BI: From 1st dose of BI or end of 10 days REP (whichever occurs later) until 2nd dose of cocktail, up to 7 days. BI+Cocktail: From 2nd dose of cocktail until last dose of BI+7 days of REP, up to 13 days.
Description: Treated set (TS): The treated set includes all subjects who signed informed consent and were treated with at least one dose of study drug.
Groups:
- Cocktail (Period 1): In period 1 (Visit 2): the cocktail reference treatment (R) consisting of 1 tablet of 0.25 milligrams (mg) of Digoxin, 0.1 milliliter (mL) oral solution of 1 mg Furosemide, 0.05 mL oral solution of 10 mg Metformin, and 1 film-coated tablet of 10 mg Rosuvastatin were taken orally, each medication as a single dose, once on Day 1 of period 1 (Visit 2).
- Cocktail+BI 730357 (Overlap Period): This group refers to the time interval where the residual effect period of the 1st dose of cocktail in period 1 overlaps with the start of the dosing of BI 730357, up to 3 days.
  3 film-coated tablets of 100 milligrams (mg) BI 730357 were taken orally twice daily (bid) with daily dose 600 mg starting from Day -7 of Visit 3.
- BI 730357 (Period 2): In period 2 (Visit 3): 3 film-coated tablets of 100 mg BI 730357 were taken orally twice daily (bid) with daily dose 600 mg from Day -7 until Day 1 of Visit 3 before the first does of combination of BI and cocktail medications (up to 7 days).
- BI 730357+Cocktail (Period 2): In period 2 (Visit 3): 3 film-coated tablets of 100 mg BI 730357 were taken orally twice daily (bid) with daily dose 600 mg from Day 1 until Day 6 of Visit 3 (7 days in total). On Day 1 of Visit 3, 1 hour after the morning dose of BI 730357, the cocktail (1 tablet of 0.25 mg of Digoxin, 0.1 mL oral solution of 1 mg Furosemide, 0.05 mL oral solution of 10 mg Metformin, and 1 film-coated tablet of 10 mg Rosuvastatin) was administered orally once.
Arm/Group | Cocktail (Period 1) | Cocktail+BI 730357 (Overlap Period) | BI 730357 (Period 2) | BI 730357+Cocktail (Period 2)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 6/15 | 1/15 | 4/15 | 4/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cocktail (Period 1) (N=15) | Cocktail+BI 730357 (Overlap Period) (N=15) | BI 730357 (Period 2) (N=15) | BI 730357+Cocktail (Period 2) (N=14)
Headache (Nervous system disorders) | 5 | 0 | 0 | 2
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Food aversion (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT04590937/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT04590937/SAP_001.pdf